CLINICAL TRIAL: NCT05551455
Title: Investigating the Endocrinological and Physiological Responses to Short-term Reduced Carbohydrate Availability in Males.
Brief Title: Endocrinological and Physiological Responses to Short-term Reduced Carbohydrate Availability in Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22/SPS/026
Record Dates: First submitted 2021-03-02; First posted 2022-09-22 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Energy Supply; Deficiency; Carbohydrate Availability
Keywords: Bone turnover markers; Testosterone; Glucose; Glycerol; Ketones; Insulin; Leptin; Ghrelin; Triglycerides; Triiodothyronine; Thyroxine; Resting Metabolic Rate (RMR); Free fatty acids; Blood pressure; ß-CTX; P1NP
MeSH Terms: conditions — Ketosis; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will complete two five-day trial-arms in randomised order, with an ~10-day washout period between interventions.
Masking Description: Masking not possible as food quantity/type will vary between interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Carbohydrate Availability (Other): Participants will complete a supervised morning cycling session daily (each morning for five days) to achieve a 15 kcal/kg FFM/day exercise energy expenditure, with samples collected pre-, during- and post-exercise. Participants will then be provided (daily) with all subsequent dietary intake for the intervention period.
  In the Normal Carbohydrate Availability trial arm, participants will be provided with 60 kcal/kg FFM/day of energy intake, to elicit a net energy availability of 45 kcal/kg FFM, with ~60% of this energy intake from carbohydrates.
  The intervention will last for four days, spanning five testing mornings (i.e. trial begins following fasted baseline assessments on morning 1, finishing with final sample collection on morning 5).
  Interventions: Other: Nutritional/dietary intake manipulation ('Normal')
- Low Carbohydrate Availability (Experimental): Participants will complete a supervised morning cycling session daily (each morning for five days) to achieve a 15 kcal/kg FFM/day exercise energy expenditure, with samples collected pre-, during- and post-exercise. Participants will then be provided (daily) with all subsequent dietary intake for the intervention period.
  In the Low Carbohydrate Availability trial arm, participants will be provided with 60 kcal/kg FFM/day of energy intake, to elicit an energy availability of 45 kcal/kg FFM, with ~1.5 g/kg provided from carbohydrate and ~70-80% of energy intake in the form of fat.
  The intervention will last for four days, spanning five testing mornings (i.e. trial begins following fasted baseline assessments on morning 1, finishing with final sample collection on morning 5).
  Interventions: Other: Nutritional/dietary intake manipulation ('Low')

INTERVENTIONS:
Other: Nutritional/dietary intake manipulation ('Normal') — Energy Intake provision (60 kcal/kg FFM/day) to elicit 'normal' energy availability (45 kcal/kg FFM/day), with 60% from carbohydrates.
  Other Names: Normal Carbohydrate Availability
  Arms: Normal Carbohydrate Availability
Other: Nutritional/dietary intake manipulation ('Low') — Energy Intake provision (60 kcal/kg FFM/day), with 1.5 g/kg of carbohydrate and 70-80% fat intake, to elicit 'low' carbohydrate availability in energy balance (45 kcal/kg FFM/day).
  Other Names: Low Carbohydrate Availability
  Arms: Low Carbohydrate Availability

SUMMARY:
Using a randomised crossover design, nine weight-stable men, aged 18 - 40 years old, will be recruited via convenience sampling from the staff and student body of LJMU and local area. Participants will be asked to follow two 4-day (~96 hours) periods of tightly controlled exercise energy expenditure (15 kcal/kg FFM/day [cycling]) and dietary intake (60 kcal/kg FFM/day) to compare a state of 'normal' energy availability (or energy balance; equivalent to 45 kcal/kg FFM/day) with concomitant 1: normal carbohydrate availability ('Normal'; ~60% of dietary intake from carbohydrate) and 2: low carbohydrate availability ('LCHF', ~1.5 g/kg carbohydrate per day, ~70 - 80% dietary intake from fat). This approximates the amount of carbohydrate consumed by an individual in a state of LEA through consuming 10 kcal/kg FFM/day with 50% of intake from carbohydrate, or ~1.5 g/kg/day of carbohydrate. In both experimental phases we will measure endocrine, metabolic and physiological parameters.

DETAILED DESCRIPTION:
Rationale:

The primary research question associated with this study is 'What is the impact of an acute period of low carbohydrate availability upon associated physiological and endocrinological markers in a cohort of healthy males?'

Extensive research has been conducted since the 1970s to determine the aetiology behind the concurrent impairment of reproductive function and low bone mineral density that is commonly observed in exercising females (De Souza et al., 2014). This research has determined that chronic low energy availability ('LEA' - the energy available from diet after energy used in exercise has been subtracted) is the key determining factor for the endocrine and physiological responses observed in the Female Athlete Triad (De Souza et al., 2014) model. However, whilst the Male Athlete Triad (Nattiv et al., 2021) and RED-S (Mountjoy et al., 2018) models identify the likely impact of LEA upon males, equivalent research identifying the physiological effects of this state in males is far behind that of females.

Moreover, whilst low energy availability has been identified as the key driver of the physiological dysregulations identified in the Female/Male Athlete Triad and RED-S models, much of the existing research has not adequately delineated between the impact of low energy availability, per se, and low carbohydrate availability. Recent research suggests that low carbohydrate availability, with or without the presence of LEA, may be a driver of the physiological dysregulations identified within the aforementioned models. For example, McKay et al (2021) have shown altered iron and immune responses and impaired exercise performance following 6-days of low carbohydrate (50 - 100 g/day) but ~normal energy availability (40 kcal•kg FFM-1•day-1), whilst no changes were apparent in a LEA (15 kcal•kg FFM-1•day-1, 60% carbohydrate) and a control group. Similarly, Heikura et al (2020) have recently shown that over 3.5 weeks, a ketogenic diet impairs markers of bone turnover compared to an energy-matched high carbohydrate diet in highly trained athletes.

Given that exercise and nutritional interventions are key for improving weight-loss and health of the general population, understanding how reduced energy and/or carbohydrate availability may affect male endocrinology and physiology is of the utmost importance. The effects and mechanisms by which low energy and/or carbohydate availability influences male physiological function therefore requires further research using well-controlled experimental research designs.

We have recently conducted a study that aimed to understand the broad physiological, endocrine and muscular responses to a period of five-days of low energy availability (analysis of samples is ongoing). The proposed study therefore now aims to extend the scope of our research to investigate the impact of four- days of low carbohydrate availability using a low-carbohydrate, high-fat diet in the presence of adequate energy availability to address this gap in the literature.

Objectives:

Primary:

To investigate the physiological responses of adult males to low carbohydrate availability whilst in energy balance over 4-days (~96 hrs, spanning five testing mornings), in contrast to an equivalent period of controlled energy balance with 'normal' carbohydrate availability in relation to muscle and endocrine parameters.

Secondary:

To investigate the wider physiological responses of adult males to low carbohydrate availability (whilst in energy balance) over 4-days (~96 hrs, spanning five testing mornings), compared to an equivalent period in controlled 'normal' carbohydrate availability in relation to whole-body physiological and metabolic status as well as body composition changes.

Study Methods:

Using a randomised cross-over design, participants will complete two interventions that will elicit conditions of 'normal' (NEA) and 'low' (LEA) carbohydrate availability whilst in energy balance, with a 10-day washout period in between conditions. Body composition changes and markers of bone turnover and reproductive health will be assessed, along with further physiological parameters.

Sample Size:

Sample size was determined based upon the primary outcome measure of Free Circulating Testosterone, the least sensitive primary outcome measures of the study.

The findings of Koehler et al (2016) were used to estimate required sample size for this study. Koehler et al (2016) reported a non-significant (P >0.05) change in Testosterone following four days of Low Energy Availability (with exercise) at 15 kcal/kg FFM/day (LEA + Ex: Pre 5.27 ± 0.46, Post 4.46 ± 0.96 ng.ml-1), compared to a control group with exercise (C + Ex: Pre 4.98 ± 0.47 Post 4.92 ± 0.53 ng.ml-1). However, a large effect size for the reduction in testosterone concentrations for LEA + Ex compared to C + Ex (d = 1.36) was observed/calculated. Therefore a post-hoc power analysis was conducted, revealing a power (1-β err probability) of 0.759 for the sample size of N = 6. To replicate these findings with greater statistical power (α err prob 0.05, 1-β err prob > 0.9) would require 8 participants, with 9 participants required to factor for a potential 10% dropout rate in participants commonly observed.

Quality:

The research plan has been reviewed internally within the research team at Liverpool John Moores University. The researcher's associated with this study and associated with the review of the study protocol are all members of staff (or a PhD Student) within the Liverpool John Moores University Research Institute for Sport & Exercise Sciences (RISES). In the 2014 RISES (LJMU) submitted 34.75 FTE (full time equivalent) to Unit of Assessment 26 (UoA26) and attained a GPA (Grade Point Average) of 3.57. Placed second on GPA in the UoA, RISES became the leading centre for Sport and Exercise Science Research Quality in the UK (4* - 61% of all activity world leading, 3* - 36% of all activity internationally excellent standard). RISES submitted the largest volume of 4* outputs (n=60) in the UoA, had 90% of the impact activity rated at 4* and had 100% of the environment rated as 4*. Importantly, out of 1,911 submissions in all 36 UoA's RISES came 11th in the entire UK for GPA achieved at REF2014, putting RISES (LJMU) amongst Oxford, UCL, LSE and Cambridge in the league tables for this metric. This makes RISES perfectly qualified to assess this research project.

ELIGIBILITY:
Inclusion Criteria:

* Gender/Sex: Male
* Age:18-40
* Healthy (as determined by pre-participation questionnaires)
* Regularly Exercising/Aerobically trained (3 + times/week, VO2max >50 ml/kg/min), as determined through participant self-identification via recruitment email/verbal communication and baseline assessment of VO2max)
* Weight-stable (within 2 kg) for the past 6-months

Exclusion Criteria:

* Gender/Sex: Female/Other
* Age - < 18 - > 40
* Health - Deemed unable to perform exercise (assessed via PAR-Q)
* Current smoker.
* Medical Condition - Those with any previous diagnosis of; Osteoporosis/low bone mineral density, cardio-vascular disease, Diabetes Mellitus, Cerebrovascular Disease, blood-related illness/disorder, Asthma or other respiratory illness/disorder, Liver Disease, Kidney Disease, gastrointestinal disease, Eating Disorder or Disordered Eating. Those currently taking prescription medication or unwell with a cold or virus at the time of participation.
* Those unwilling to adhere to the study's methodological requirements (including adhering to alterations in diet and training - inc. alcohol abstention) from the day prior to intervention onset (24 hrs pre-intervention) to completion of follow-up assessments (day 5).
* Those following a restrictive diet (e.g. vegans)
* Those with food allergies and/or food intolerances
* Training status - Does not train 3 + times/week (over past 6 months on average) and/or have a VO2max >50 ml/kg/min.
* Any athletes that may be tested for substances on the WADA banned substances list

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in blood bone turnover markers: ß-CTX (Bone Resorption) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes in blood-borne bone (re)modelling marker ß-CTX (Bone Resorption) following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood bone turnover markers: P1NP (Bone Formation) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes in blood-borne bone (re)modelling marker P1NP (Bone Formation)
Changes in blood metabolites/hormones: Testosterone | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating testosterone concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability

SECONDARY OUTCOMES:
Change in resting substrate utilisation | Days 1, 3 and 5 of each intervention
  Analysis of changes in resting substrate utilisation. Assessed using indirect calorimetry.
Changes in sub-maximal Exercise Energy Expenditure | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes in sub-max exercise energy expenditure and substrate utilisation at standardised exercise intensities. Assessed using indirect calorimetry.
Changes in sub-maximal exercise substrate utilisation | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes in sub-max exercise energy expenditure and substrate utilisation at standardised exercise intensities. Assessed using indirect calorimetry.
Immune function | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to saliva-based markers of immune function
Changes in Initial Orthostatic Hypotension (IOH) | Pre- and post-intervention (days 1 and 5) for both intervention
  Analysis of changes in IOH, assessed via blood pressure finometry and questionnaire
Change in Profile of Mood States | Pre- and post-intervention (days 1 and 5) per intervention
  Analysis of changes in Psychological/mood, assessed via the POMS-40 questionnaire
Change in subjective hunger | Days 1, 2, 3, 4 & 5 per intervention
  Analsis of changes in subjective hunger, assessed via visual analogue scales
Change in sexual drive/libido | Pre- and post-intervention (days 1 and 5)
  Analysis of subjective sex-drive/libido changes, assessed via visual analogue scale
Physical activity energy expenditure (PAEE) | Continuous monitoring during intervention period (5-days)
  Analysis of PAEE alterations, assessed via wrist-worn accelerometers (acti-watch)
Sleep duration and quality | Continuous monitoring during intervention period (5-days)
  Analysis of sleep alterations, assessed via wrist-worn device and sleep diary (collectively quantified by analysis of sleep duration, sleep latency, time of sleep onset, no of wakes during night, subjective sleep quality visual analogue scale)
Changes in Body Composition: Body Mass (kg) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Body Mass Index (kg/m^2) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Fat Mass (kg) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Body Fat Percentage (%) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Fat Free Mass (kg) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Skeletal Muscle Mass (kg) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Total Body Water (l) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Total Body Water (%) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Extra-cellular Water (l) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Extra-cellular Water (%) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in Body Composition: Extra-cellular Water/Total Body Water ratio | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of body composition changes - assessed using bio-electrical impedance analysis (BIA)
Changes in blood metabolites/hormones: Ketones | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating ketones concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: Glucose | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating glucose concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: Free fatty Acids | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating free fatty acid concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: Insulin | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating insulin concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: Cortisol | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating cortisol concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: HDL | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating HDL concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: LDL | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating LDL concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: glycerol | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating glycerol concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: Leptin | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating Leptin concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: IGF-1 | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating IGF-1 concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Alterations to skeletal muscle glycogen | Days 1 & 5 per intervention (pre-post)
  Assessment of alterations in skeletal muscle glycogen content
Alterations to Intra-muscular lipid profile: lipid droplet content | Days 1 & 5 per intervention (pre-post)
  Assessment of alterations in lipid droplet content
Alterations to Intra-muscular lipid profile: lipid droplet morphology | Days 1 & 5 per intervention (pre-post)
  Assessment of alterations in lipid droplet morphology
Alterations to Intra-muscular lipid profile: lipid droplet associated proteins | Days 1 & 5 per intervention (pre-post)
  Assessment of alterations in lipid droplet associated proteins
Resting Metabolic Rate | Days 1, 3 and 5 of each intervention
  Analysis of changes to Resting Metabolic Rate (kcal/day) following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability
Changes in blood metabolites/hormones: Triiodothyronine (T3) | Days 1, 2, 3, 4 & 5 per intervention
  Analysis of changes to circulating T3 concentrations following short term energy balance with a) normal carbohydrate availability and b) low carbohydrate availability

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Areta, Study Director — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No